CLINICAL TRIAL: NCT04622501
Title: Spinal Epidural Lipomatosis: a Case Report and Review of the Literature
Status: Completed | Type: Observational
Sponsor: Canadian Memorial Chiropractic College (Other)
Responsible Party: Sponsor
Other Study IDs: 202015
Record Dates: First submitted 2020-08-10; First posted 2020-11-10 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: posterior spinal decompression and posterior spinal instrumented fusion — posterior spinal decompression and posterior spinal instrumented fusion performed on a patient with Spinal Epidural Lipomatosis

SUMMARY:
Introduction Lumbar spinal epidural lipomatosis (SEL) is a rare condition defined by an excessive deposition of adipose tissue in the lumbar spinal canal. The objective of this case report is to document a clinical case of SEL presenting within a multidisciplinary spine clinic and to compare our clinical findings and management with the current literature.

Case presentation A 51-year-old female presented at a spine clinic with low back pain, bilateral leg pain and difficulty walking. MR imaging of the lumbar spine showed L4-L5 and L5-S1 degenerative disk disease with evidence of severe central canal stenosis due to extensive epidural lipomatosis. The patient was initially advised to lose weight, undergo a course of physiotherapy, and consult with the pain clinic. Because of lack of improvement, the patient was scheduled for L4-S1 posterior spinal decompression and L4-L5 posterior spinal instrumented fusion.

Discussion The discussion will include the diagnosis of SEL, imaging appearance, its risk factors, etiology and management.

Conclusion This case report describes a case of lumbar spinal stenosis due to SEL with neurological symptoms. Some risk factors have also been identified in the literature. MRI is considered as the reference standard for its diagnosis. The therapeutic approach of patients with SEL is not standardized. Thus, reporting and investigating the diagnostic process and treatment of this patient will positively contribute to better management for other future patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults patient with a clinical diagnosis of Spinal Epidural Lipomatosis (MRI and clinical diagnosis)

Exclusion Criteria:

* Absence of clinical diagnosis of Spinal Epidural Lipomatosis

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients consulting in a multidisciplinary spine clinic
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Low back pain | 3 months before surgery
  Visual Pain Scale (0-10)
Low back pain | 6 weeks after surgery
  Visual Pain Scale (0-10)
Distance Walking | 3 months before surgery
  Distance walking (meter)
Distance Walking | 6 weeks after surgery
  Distance walking (meter)
Low back pain | 3 months after surgery
  Visual Pain Scale (0-10)
Low back pain | 1 year after surgery
  Visual Pain Scale (0-10)
Distance walking | 3 months after surgery
  Distance walking (meter)
Distance walking | 1 year after surgery
  Distance walking (meter)

CONTACTS AND LOCATIONS:
Locations (1):
- CMCC, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Borre DG, Borre GE, Aude F, Palmieri GN. Lumbosacral epidural lipomatosis: MRI grading. Eur Radiol. 2003 Jul;13(7):1709-21. doi: 10.1007/s00330-002-1716-4. Epub 2002 Dec 13. PMID 12835988
- [Background] Fogel GR, Cunningham PY 3rd, Esses SI. Spinal epidural lipomatosis: case reports, literature review and meta-analysis. Spine J. 2005 Mar-Apr;5(2):202-11. doi: 10.1016/j.spinee.2004.05.252. PMID 15795966
- [Background] Agha RA, Borrelli MR, Farwana R, Koshy K, Fowler AJ, Orgill DP; SCARE Group. The SCARE 2018 statement: Updating consensus Surgical CAse REport (SCARE) guidelines. Int J Surg. 2018 Dec;60:132-136. doi: 10.1016/j.ijsu.2018.10.028. Epub 2018 Oct 18. PMID 30342279
- [Background] Fassett DR, Schmidt MH. Spinal epidural lipomatosis: a review of its causes and recommendations for treatment. Neurosurg Focus. 2004 Apr 15;16(4):E11. PMID 15191340
- [Background] Theyskens NC, Paulino Pereira NR, Janssen SJ, Bono CM, Schwab JH, Cha TD. The prevalence of spinal epidural lipomatosis on magnetic resonance imaging. Spine J. 2017 Jul;17(7):969-976. doi: 10.1016/j.spinee.2017.02.010. Epub 2017 Mar 3. PMID 28263890
- [Background] Yildirim B, Puvanesarajah V, An HS, Novicoff WM, Jain A, Shen FH, Hassanzadeh H. Lumbosacral Epidural Lipomatosis: A Retrospective Matched Case-Control Database Study. World Neurosurg. 2016 Dec;96:209-214. doi: 10.1016/j.wneu.2016.08.125. Epub 2016 Sep 5. PMID 27609448
- [Background] Kim K, Mendelis J, Cho W. Spinal Epidural Lipomatosis: A Review of Pathogenesis, Characteristics, Clinical Presentation, and Management. Global Spine J. 2019 Sep;9(6):658-665. doi: 10.1177/2192568218793617. Epub 2018 Aug 13. PMID 31448201
- [Background] Malone JB, Bevan PJ, Lewis TJ, Nelson AD, Blaty DE, Kahan ME. Incidence of spinal epidural lipomatosis in patients with spinal stenosis. J Orthop. 2017 Nov 6;15(1):36-39. doi: 10.1016/j.jor.2017.11.001. eCollection 2018 Mar. PMID 29203971
- [Background] Walchli B, Benini A. Spinal epidural lipomatosis. Swiss Med Wkly. 2001 Jun 16;131(23-24):359. doi: 10.4414/smw.2001.09739. No abstract available. PMID 11486570
- [Background] Ferlic PW, Mannion AF, Jeszenszky D, Porchet F, Fekete TF, Kleinstuck F, Haschtmann D. Patient-reported outcome of surgical treatment for lumbar spinal epidural lipomatosis. Spine J. 2016 Nov;16(11):1333-1341. doi: 10.1016/j.spinee.2016.06.022. Epub 2016 Jun 27. PMID 27363757